CLINICAL TRIAL: NCT05094713
Title: Effects of Tissue Flossing on Muscle Contractile Properties and Jumping Performance in Recreationally Active Students
Brief Title: Effects of Muscle Flossing on Quadriceps Muscle Potentiation
Acronym: MF_TMG_CMJ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Science and Research Centre Koper (Other)
Collaborators: University of Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: MFPAP
Record Dates: First submitted 2021-10-13; First posted 2021-10-26 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Ischemia; Placebo - Control
Keywords: tissue flossing
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Intervention Model Description: Crossover randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flossing - control (Other): Control group where flossing wrapping pressure is between 20 and 30 mmHg
  Interventions: Other: Low wrapping pressure
- Flossing with medium wrapping pressure (Experimental): A flossing band will be applied over tight musculature with medium wrapping pressure
  Interventions: Other: Flossing experimental group

INTERVENTIONS:
Other: Flossing experimental group — Flossing of the tight muscles with medium wrapping pressure, which is individualized in based on the tight circumference of the participant.
  Other Names: Muscle flossing
  Arms: Flossing with medium wrapping pressure
Other: Low wrapping pressure — Control group where flossing wrapping pressure is between 20 and 30 mmHg
  Other Names: CONTROL
  Arms: Flossing - control

SUMMARY:
Tissue flossing involves wrapping a thick rubber band around a joint or muscle, which can partially occlude blood flow. In practice, it is often used while concomitantly performing a range of motion exercises (ROM) for 1 to 3 minutes in duration. The mechanisms involved in tissue flossing with a floss band may be similar to those involved in ischemic preconditioning. Previous results would support the use of tissue flossing on ROM, while there are no clear conclusions on post-activation effects on sports-related performance and muscle contractile properties. This may be attributed to the different methodologies used in the studies. Therefore, the time course associated with tissue flossing benefits remains to be investigated.

DETAILED DESCRIPTION:
Nowadays, various methods are used for acute performance enhancement. The most recent of these is tissue flossing, which is becoming increasingly popular for both performance enhancement and rehabilitation. However, the effects of flossing on athletic performance have not been clearly demonstrated, which could be due to differences in the methodology used. In particular, the rest periods between the end of the preconditioning activity and the performance of the criterion task or assessment tools varied considerably in the published literature. Therefore, the present study aimed to investigate the effects of applying tissue flossing to the thigh on bilateral countermovement jump performance and contractile properties of vastus lateralis (VL) muscle. Nineteen recreational athletes (11 males; aged 23.1 ± 2.7 years) were randomly assigned to days of flossing application (3 sets for 2 min of flossing with 2 min rest between sets) with preset experimental pressure (EXP = 95 ± 17.4 mmHg) or control condition (CON = 18.9 ± 3.5 mmHg). The first part of the measurements was performed before and after warm-up consisting of 5 min of cycling followed by dynamic stretching and specific jumping exercises, while the second part consisted of six measurement points after flossing application (0.5, 3, 6, 9, 12, 15 min).

ELIGIBILITY:
Inclusion Criteria:

* Healthy and physically active individuals
* without a history of lower limb injuries and/or surgeries at least 1 year prior to investigation.

Exclusion Criteria:

* neuromuscular and metabolic disorders;
* the presence of acute and/or chronic pain
* alcohol and drug consumption etc.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Contractile muscle properties | 75 min
  Contractile muscle properties assessed using tensiomyography (Tc, Dm, Tr, Ts, Td)

SECONDARY OUTCOMES:
CMJ jump height | 75 min
  Counter-movement jump height assessed using force plate

OTHER OUTCOMES:
Rate of perceived exertion | 75 min
  Rate of perceived exertion of fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Armin Paravlic, PhD, Principal Investigator — SRC Koper and Faculty of Sport
Locations (1):
- Science and Research centre Koper, Koper, Slovenia

REFERENCES:
- [Result] Paravlic AH, Segula J, Drole K, Hadzic V, Pajek M, Vodicar J. Tissue Flossing Around the Thigh Does Not Provide Acute Enhancement of Neuromuscular Function. Front Physiol. 2022 Apr 27;13:870498. doi: 10.3389/fphys.2022.870498. eCollection 2022. PMID 35574482
- See also: Published article — https://www.frontiersin.org/articles/10.3389/fphys.2022.870498/full